CLINICAL TRIAL: NCT00941070
Title: A Phase 2 Study of Triapine® (NSC #663249) and Cisplatin in Combination With Pelvic Radiation for Treatment of Stage IB2-IVa Cervical Cancer or Stage II-IV Vaginal Cancer
Brief Title: Triapine, Cisplatin, and Radiation Therapy in Treating Patients With Cervical Cancer or Vaginal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02896; NCI-2012-02896 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000647544; CASE 11808 (Other: Case Comprehensive Cancer Center); 8327 (Other: CTEP); P30CA043703 (NIH); U01CA062502 (NIH)
Record Dates: First submitted 2009-07-16; First posted 2009-07-17 (Estimated); Results first posted 2013-05-13 (Estimated); Last update posted 2017-11-17 (Actual); Status verified 2017-10

CONDITIONS: Recurrent Cervical Cancer; Recurrent Vaginal Cancer; Stage IB Cervical Cancer; Stage II Vaginal Cancer; Stage IIA Cervical Cancer; Stage IIB Cervical Cancer; Stage III Cervical Cancer; Stage III Vaginal Cancer; Stage IVA Cervical Cancer; Stage IVA Vaginal Cancer; Stage IVB Cervical Cancer; Stage IVB Vaginal Cancer; Therapy-related Toxicity
MeSH Terms: conditions — Uterine Cervical Neoplasms; Vaginal Neoplasms | interventions — 3-aminopyridine-2-carboxaldehyde thiosemicarbazone; Cisplatin; Fluorodeoxyglucose F18; Magnetic Resonance Spectroscopy; 2-phenyl-6-(2'-(4'-(ethoxycarbonyl)thiazolyl))thiazolo(3,2-b)(1,2,4)triazole

ARMS (1):
- Treatment (cisplatin, triapine, radiation therapy) (Experimental): Patients receive cisplatin IV over 90 minutes on days 2, 9, 16, 23, and 30 and triapine IV on days 1, 3, 5, 8, 10, 12, 15, 17, 19, 22, 24, 26, 29, 31, and 33. Patients also undergo pelvic external beam radiotherapy 5 days a week during weeks 1-5. Patients may undergo parametrial boost radiation and intracavitary low-dose or high-dose rate brachytherapy as clinically indicated.
  Patients undergo whole-body F-18 fluorodeoxyglucose-PET/CT imaging at baseline, at 3 months after completion of study treatment, and at disease progression. Patients complete Sexual Function-Vaginal Changes Questionnaire and a smoking behavior questionnaire at baseline, at 3 months after completion of study treatment, and at disease progression.
  Interventions: Drug: triapine; Drug: cisplatin; Radiation: external beam radiation therapy; Procedure: quality-of-life assessment; Other: questionnaire administration; Radiation: fludeoxyglucose F 18; Procedure: positron emission tomography; Procedure: computed tomography

INTERVENTIONS:
Drug: triapine — Given IV
  Other Names: 3-AP; OCX-191
Drug: cisplatin — Given IV
  Other Names: CACP; CDDP; CPDD; DDP
Radiation: external beam radiation therapy — Undergo pelvic external beam radiation therapy
  Other Names: EBRT
Procedure: quality-of-life assessment — Ancillary studies
  Other Names: quality of life assessment
Other: questionnaire administration — Ancillary studies
Radiation: fludeoxyglucose F 18 — Undergo FDG-PET/CT
  Other Names: 18FDG; FDG
Procedure: positron emission tomography — Undergo FDG-PET/CT
  Other Names: FDG-PET; PET; PET scan; tomography, emission computed
Procedure: computed tomography — Undergo FDG-PET/CT
  Other Names: tomography, computed

SUMMARY:
This phase II trial is studying how triapine and cisplatin given together with radiation therapy works in treating patients with cervical cancer or vaginal cancer. Triapine may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Radiation therapy uses high-energy x-rays to kill tumor cells. Giving triapine together with cisplatin may make tumor cells more sensitive to radiation therapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine three-month fasting F-18 fluorodeoxyglucose (FDG) positron emission tomography (PET/CT) imaging complete metabolic response as defined by the European Organization for Research and Treatment of Cancer (EORTC) PET study group.

SECONDARY OBJECTIVES:

I. To determine 6-month progression-free survival rate as calculated from the date of first treatment until date of disease progression, relapse, or death.

II. To quantitate change in pre-treatment standard uptake value (SUV) on PET/CT and post-treatment PET/CT or disease progression PET/CT.

III. To quantitate pre-treatment, during treatment and 3-mo post-treatment grade 2 or higher gastrointestinal, genitourinary, and sexual function toxicity resulting from Triapine®, cisplatin, and radiation therapy as measured by CTCAE v3.0, which will be utilized until December 31, 2010; CTCAE v4.0 will be utilized beginning January 1, 2011.

IV. To associate smoking habit (non-smoker, smoker who quit during therapy, smoker) with 3-mo post-treatment PET/CT metabolic response and 3-mo best overall clinical response as measured by RECIST criteria after Triapine®, cisplatin, and radiation therapy.

V. To associate HPV or non-HPV sub-type cervical cancer with 3-mo post-treatment PET/CT metabolic response and 3-mo best overall clinical response as measured by RECIST criteria after Triapine®, cisplatin, and radiation therapy.

OUTLINE: This is a multicenter study. Patients are stratified according to brachytherapy treatment (planned intracavitary brachytherapy vs none).

Patients receive cisplatin IV over 90 minutes on days 2, 9, 16, 23, and 30 and triapine IV on days 1, 3, 5, 8, 10, 12, 15, 17, 19, 22, 24, 26, 29, 31, and 33. Patients also undergo pelvic external beam radiotherapy 5 days a week during weeks 1-5. Patients may undergo parametrial boost radiation and intracavitary low-dose or high-dose rate brachytherapy as clinically indicated.

Patients undergo whole-body F-18 fluorodeoxyglucose-PET/CT imaging at baseline, at 3 months after completion of study treatment, and at disease progression. Patients complete Sexual Function-Vaginal Changes Questionnaire and a smoking behavior questionnaire at baseline, at 3 months after completion of study treatment, and at disease progression.

After completion of study treatment, patients are followed periodically for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Female patients must have histologically confirmed (tumor tissue biopsy) primary clinical stage IB2-IVB cervical cancer or clinical stage II-IVB vaginal cancer not amenable to curative surgical resection alone to be eligible; patients with stage IVB cervical cancer may receive systemic chemotherapy for treatment of metastatic disease a) after the 3-month post-therapy PET scan and b) if the 3-month post-therapy PET scan documents progressive disease at the discretion of the treating physician
* Patients with other active invasive malignancies are excluded; patients with prior malignancies (except non-melanoma skin cancer or prior in situ carcinoma of the cervix, patients with synchronous or past history of primary endometrial cancer meeting all conditions of a) stage not greater than IB, b) no more than superficial myometrial invasion, c) without vascular or lymphatic invasion, and d) no poorly differentiated subtypes including papillary serous, clear cell or other FIGO grade 3 lesions; patients with other invasive malignancies who had (or have) cancer present within the last five years are excluded; patients are excluded if they have received prior low abdominal or pelvic radiotherapy for any reason that would contribute radiation dose that would exceed tolerance of normal tissues
* Life expectancy of greater than 3 months
* Absolute neutrophil count >= 1,500/uL
* Platelets >= 100,000/uL
* Hemoglobin >= 10 g/dL
* Total bilirubin =< 2.0 mg/dL
* AST(SGOT)/ALT(SGPT) =< 2.5 X institutional upper limit of normal
* PT/aPTT =< 1.5 X institutional upper limit of normal
* Patients should have a serum creatinine =< 1.5mg/dL to receive weekly intravenous cisplatin chemotherapy

  * Patients whose serum creatinine is between 1.5 and 1.9 mg/dL are eligible for cisplatin chemotherapy if the estimated creatinine clearance is >= 30 ml/min; patients eligible for cisplatin chemotherapy using the criteria for creatinine clearance may also receive intravenous Triapine®
* Women of child-bearing potential and male partners must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Patients must demonstrate ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier are excluded
* Patients may not be receiving any other investigational agents
* Patients with known brain metastases should be excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurological dysfunction that would confound the evaluation of neurological and other adverse events
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to Triapine® or other agents used in study
* Patients unable to receive intravenous chemotherapies as a consequence of poor vascular access are ineligible
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, known inadequately controlled hypertension, significant pulmonary disease including dyspnea at rest, patients requiring supplemental oxygen, or poor pulmonary reserve; proteinuria or clinically significant renal function impairment (baseline serum creatinine > 2mg/dL), or psychiatric illness/social situations that would limit compliance with study requirements are excluded
* Patients with known glucose-6-phosphate dehydrogenase deficiency (G6PD) are excluded as the antidote methylene blue for Triapine® toxicity may be at best ineffective in such patients and may have the potential to complicate the clinical situation by provoking hemolysis
* Pregnant women are excluded from this study because Triapine® is a heterocyclic carboxaldehyde thiosemicarbazone with the potential for teratogenic or abortifacient effects; screening beta-hcg levels and diagnostic tests will be used to determine eligibility; because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with Triapine®, breastfeeding should be discontinued if the mother is treated with Triapine®; these potential risks may also apply to other agents used in this study
* Patients not willing to agree to use appropriate contraception while on trial will be excluded
* HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with Triapine®; in addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy; appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated; HIV testing is not mandatory; patients that are known to be HIV-positive are ineligible if they are receiving combination antiretroviral therapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2009-07; Primary Completion 2012-04 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles Kunos, Principal Investigator — Case Comprehensive Cancer Center
Locations (1):
- Case Western Reserve University, Cleveland, Ohio, United States

REFERENCES:
- [Derived] Yun T, Liu Z, Wang J, Wang R, Zhu L, Zhu Z, Wang X. Microenvironment immune response induced by tumor ferroptosis-the application of nanomedicine. Front Oncol. 2022 Sep 16;12:1019654. doi: 10.3389/fonc.2022.1019654. eCollection 2022. PMID 36185311
- [Derived] Chao J, Synold TW, Morgan RJ Jr, Kunos C, Longmate J, Lenz HJ, Lim D, Shibata S, Chung V, Stoller RG, Belani CP, Gandara DR, McNamara M, Gitlitz BJ, Lau DH, Ramalingam SS, Davies A, Espinoza-Delgado I, Newman EM, Yen Y. A phase I and pharmacokinetic study of oral 3-aminopyridine-2-carboxaldehyde thiosemicarbazone (3-AP, NSC #663249) in the treatment of advanced-stage solid cancers: a California Cancer Consortium Study. Cancer Chemother Pharmacol. 2012 Mar;69(3):835-43. doi: 10.1007/s00280-011-1779-5. Epub 2011 Nov 22. PMID 22105720

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from local medical clinic from July 2009 through November 2011
Period: Overall Study
Arm/Group | Treatment (Cisplatin, Triapine, Radiation Therapy)
Started | 26
Completed | 25
Not Completed | 1
Not completed — Patient non-compliant | 1

BASELINE CHARACTERISTICS:
Population: Baseline demographic characteristics include all 26 patients. Study specific characteristics only include the 25 patients that received treatment.
Arm/Group | Treatment (Cisplatin, Triapine, Radiation Therapy)
Number analyzed (Participants) | 26
Age, Customized [Number; unit: participants]
  30-39 | 1
  40-49 | 7
  50-59 | 11
  60-69 | 6
  70-79 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 24
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 18
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 26
GOG Performance Status [Number; unit: participants] — One patient was non-compliant and received no therapy. Patient was excluded from study specific baseline characteristics. The Gynecologic Oncology Group (GOG) performance status reflects individual daily living activities on a scale of 0 (fully active with symptoms) to 5 (dead).
  participants
    0 | 23
    1 | 2
Histopathology [Number; unit: participants] — One patient was non-compliant and received no therapy. Patient was excluded from study specific baseline characteristics.
  participants
    Squamous cell carcinoma | 23
    Adenosquamous carcinoma | 1
    Adenocarcinoma | 1
Tumor Grade [Number; unit: participants] — One patient was non-compliant and received no therapy. Patient was excluded from study specific baseline characteristics.
  participants
    Grade 2 | 13
    Grade 3 | 12
Cervical Stromal Invasion [Number; unit: participants] — One patient was non-compliant and received no therapy. Patient was excluded from study specific baseline characteristics.
  participants
    Less than 2/3rds invasion | 3
    2/3rds or greater invasion | 22
Lymphovascular invasion [Number; unit: participants] — One patient was non-compliant and received no therapy. Patient was excluded from study specific baseline characteristics.
  participants
    Absent | 7
    Present | 18
International Federation of Gynecology and Obstetrics (FIGO) Stage [Number; unit: participants] — One patient was non-compliant and received no therapy. Patient was excluded from study specific baseline characteristics.
  participants
    Cervix IB2 Node Negative | 1
    Cervix IB2 Node Positive | 4
    Cervix IIA | 4
    Cervix IIB | 1
    Cervix IIIB | 10
    Cervix IVB | 2
    Vagina II | 2
    Vagina IVA | 1
HPV Genotyping [Number; unit: participants] — Cervical cancer genotyping
  participants
    HPV 16 | 15
    HPV 18 | 4
    HPV-naive | 6

OUTCOME MEASURES:

1. Primary Outcome: Fasting F-18 Fluorodeoxyglucose (FDG) Positron Emission Tomography (PET/CT) Imaging Complete Metabolic Response, Reported Following National Cancer Institute (NCI) and European Organization for Research and Treatment of Cancer (EORTC) Guidelines.
Description: To quantitate change in pre-treatment standard uptake value (SUV) on PET/CT and posttreatment PET/CT or disease progression PET/CT. Change in PET/CT SUV will be associated with 3-month best overall clinical response.
Time Frame: post therapy at 3 months
Population: 1 patient was non-compliant and received no therapy. Pt was excluded from analyses. 1 patient died from an unrelated health event after completing radiation and experimental chemotherapy and did not undergo 3-month F-18 FDG study.
Measure: Median (Inter-Quartile Range); unit: Standard uptake value (SUV)
Arm/Group | Treatment (Cisplatin, Triapine, Radiation Therapy)
Number analyzed (Participants) | 24
Standard uptake value (SUV)
  Pretherapy SUV | 14.6 [12.1 to 17.7]
  Posttherapy SUV | 2.6 [2.0 to 3.4]

2. Secondary Outcome: Clinical and Objective Response Assignment
Description: Number of patients with a complete clinical responses defined as disappearance of all target lesions. A complete metabolic response on PET/CT will be defined as absence of abnormal FDG uptake at sites of abnormal FDG uptake noted on pre-treatment FDG-PET study.
Time Frame: post therapy at 3 months
Population: Patients that completed the 3-month F-18 FDG study.
Measure: Number; unit: participants
Arm/Group | Treatment (Cisplatin, Triapine, Radiation Therapy)
Number analyzed (Participants) | 25
participants | 21

3. Secondary Outcome: Clinical and Objective Response Assignment
Description: as for outcome 2
Time Frame: one month follow up assessment
Population: Patients that completed the the 3-month 18F-FDG PET/CT. One patient died from an unrelated health event after completing radiation and experimental chemotherapy and was excluded from analyse.
Measure: Number; unit: participants
Arm/Group | Treatment (Cisplatin, Triapine, Radiation Therapy)
Number analyzed (Participants) | 24
participants | 23

4. Secondary Outcome: Clinical and Objective Response Assignment
Description: as for outcome 2
Time Frame: three month follow up assessment
Population: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Treatment (Cisplatin, Triapine, Radiation Therapy)
Number analyzed (Participants) | 24
participants | 23

5. Secondary Outcome: Percent of Patients With Incidence of Grade 2 or Higher Gastrointestinal and Genitourinary Toxicity, Assessed Using CTCAE v3.0 Until December 31, 2010 and CTCAE v4.0 Beginning January 1, 2011
Description: Information will include the type, severity, time of onset, time of resolution, and the probable association with the study regimen. Frequency tables will be constructed to summarize observed incidence by severity and type of toxicity.
Time Frame: After 5 weeks of radiation therapy
Population: All patients who receive at least one dose of Triapine® and cisplatin treatment.
Measure: Number; unit: percentage of patients
Arm/Group | Treatment (Cisplatin, Triapine, Radiation Therapy)
Number analyzed (Participants) | 25
percentage of patients | 0

6. Secondary Outcome: Progression-free Survival
Description: Percentage of patients that did not have disease progression. Estimates of progression-free survival will be computed using the product-limit estimate of Kaplan and Meier.
Time Frame: at 18 months from study entry
Population: Patients that completed the the 3-month 18F-FDG PET/CT.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Treatment (Cisplatin, Triapine, Radiation Therapy)
Number analyzed (Participants) | 25
percentage of patients | 67 [56 to 78]

7. Secondary Outcome: PET/CT Scan Metabolic Activity
Description: Descriptive tabular data reporting mean, standard deviation, minimum, maximum provided by metabolic response cohort. Status of 3-month post-treatment metabolic response associated with clinical response measured by RECIST criteria and with overall clinical outcome. Kaplan-Meier (product-limit) method of survival estimation used. Tests of equivalence of the estimates compared using the Wilcoxon long-rank test using P 0.05. Cox proportional hazards regression models used in multivariate analyses.
Time Frame: Baseline (pre-therapy)
Population: Patients that completed the 3-month 18F-FDG PET/CT
Measure: Median (Inter-Quartile Range); unit: Standard Uptake Value (SUV)
Arm/Group | Treatment (Cisplatin, Triapine, Radiation Therapy)
Number analyzed (Participants) | 25
Standard Uptake Value (SUV) | 14.6 [12.1 to 17.7]

8. Secondary Outcome: PET/CT Scan Metabolic Activity
Description: as for outcome 7
Time Frame: 3 months post-treatment
Population: Patients that completed 3-month 18F-FDG PET/CT
Measure: Median (Inter-Quartile Range); unit: Standard Uptake Value (SUV)
Arm/Group | Treatment (Cisplatin, Triapine, Radiation Therapy)
Number analyzed (Participants) | 24
Standard Uptake Value (SUV) | 2.6 [2.0 to 3.4]

9. Secondary Outcome: PET/CT Scan Metabolic Activity
Description: as for outcome 7
Time Frame: Up to 5 years
Population: Data were not collected as the study was terminated prior to the time period for collection.
Groups:
- Treatment (Cisplatin, Triapine, Radiation Therapy): Patients receive cisplatin and undergo pelvic external beam radiotherapy 5 days a week during weeks 1-5. Patients may undergo parametrial boost radiation and intracavitary low-dose or high-dose rate brachytherapy as clinically indicated.
  Patients undergo whole-body F-18 fluorodeoxyglucose-PET/CT imaging at baseline, at 3 months after completion of study treatment, and at disease progression.
Arm/Group | Treatment (Cisplatin, Triapine, Radiation Therapy)
Number analyzed (Participants) | 0

10. Secondary Outcome: Change in Sexual Function, Assessed Using the Sexual Function-Vaginal Changes Questionnaire
Time Frame: Baseline to up to 5 years
Population: Data were not collected as the study was terminated prior to the time period for collection.
Groups:
- Treatment (Cisplatin, Triapine, Radiation Therapy): Patients receive cisplatin and undergo pelvic external beam radiotherapy 5 days a week during weeks 1-5. Patients may undergo parametrial boost radiation and intracavitary low-dose or high-dose rate brachytherapy as clinically indicated.
  Patients undergo whole-body F-18 fluorodeoxyglucose-PET/CT imaging at baseline, at 3 months after completion of study treatment, and at disease progression. Patients complete Sexual Function-Vaginal Changes Questionnaire and a smoking behavior questionnaire at baseline, at 3 months after completion of study treatment, and at disease progression.
Arm/Group | Treatment (Cisplatin, Triapine, Radiation Therapy)
Number analyzed (Participants) | 0

11. Secondary Outcome: Change in Smoking Behavior, Assessed Using the Smoking Questionnaire and Cessation Counseling
Time Frame: 18 months from study entry
Measure: Number; unit: participants
Arm/Group | Treatment (Cisplatin, Triapine, Radiation Therapy)
Number analyzed (Participants) | 25
participants
  Non-Smokers | 9
  Smokers that quit while on study | 11
  Current smokers | 5

12. Secondary Outcome: Progression Free Survival by HPV Subtype
Description: Tabular descriptive data will be presented. HPV sub-type will be associated with treatment related toxicity, clinical response, PET metabolic response, and overall clinical outcome. Kaplan-Meier (product-limit) method of survival estimation will be used. Tests of equivalence of the estimates will be compared using the Wilcoxon long-rank test using a threshold for statistical significance of P 0.05. Cox proportional hazards regression models will be used in multivariate analyses.
Time Frame: Baseline
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Treatment (Cisplatin, Triapine, Radiation Therapy)
Number analyzed (Participants) | 25
percentage of patients
  HPV16/18 | 74 [63 to 85]
  HPV-naive tumors | 83 [62 to 98]

13. Post Hoc Outcome: Progression Free Survival by Smoking Status
Description: Percent of patients that were progression free by smoking status
Time Frame: at 18 months from study entry
Measure: Number (95% Confidence Interval); unit: percentage of paticipants
Arm/Group | Treatment (Cisplatin, Triapine, Radiation Therapy)
Number analyzed (Participants) | 25
percentage of paticipants
  Non-Smokers | 76 [62 to 90]
  Smokers that quit while on study | 89 [79 to 99]
  Smokers | 50 [25 to 75]

ADVERSE EVENTS:
Time Frame: Adverse events were collected while patients were on treatment through the 6 month follow up visit. This occurred over a 3 year period that patients were on study.
Arm/Group | Treatment (Cisplatin, Triapine, Radiation Therapy)
Serious Adverse Events (participants affected / at risk) | 9/25
Other Adverse Events (participants affected / at risk) | 25/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Cisplatin, Triapine, Radiation Therapy) (N=25)
Abdominal pain (Gastrointestinal disorders) | 1
Alanine transaminase (ALT) increased (Investigations) | 1
Anemia (Blood and lymphatic system disorders) | 1
Aspartate aminotransferase (AST) increased (Investigations) | 1
Cardiac arrythmia- Atrial Fibrillation (Cardiac disorders) | 1
Deep Vein Thrombosis (Vascular disorders) | 2
Elevated alkaline phosphatase (Investigations) | 1
Hypernatremia (Metabolism and nutrition disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 1
Hypochloride (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 4
Hypomagnesemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Hypotension (Vascular disorders) | 1
INR-international normalized ratio increased (Investigations) | 1
Leukocytopenia-white blood cell decrease (Investigations) | 1
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 — Mallory-Weiss Tears
Mallory Weiss tears-upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Stroke (Nervous system disorders) | 1
Thrombocytopenia-Platelet count decreased (Investigations) | 2
Thromboembolic event (Vascular disorders) | 1
Urinary tract infection (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Cisplatin, Triapine, Radiation Therapy) (N=25)
Abdominal pain (Gastrointestinal disorders) | 3
Alanine transaminase (ALT) increased (Investigations) | 6
Alkaline phosphatase increased (Investigations) | 3
Anemia (Blood and lymphatic system disorders) | 24
Anorexia (Metabolism and nutrition disorders) | 3
Aspartate aminotransferase (AST) increased (Investigations) | 3
Chest Pain (non-cardiac) (General disorders) | 2
Constipation (Gastrointestinal disorders) | 10
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Depression (Psychiatric disorders) | 2
Diarrhea (Gastrointestinal disorders) | 14
Dizziness (Nervous system disorders) | 2
Dysgeusia (Nervous system disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4
Elevated GGT (gamma-Glutamyl transpeptidase) (Investigations) | 6
Elevated Lactate dehydrogenase (LDH) (Metabolism and nutrition disorders) | 3
Elevated creatinine (Investigations) | 3
Fatigue (General disorders) | 11
Fever (General disorders) | 3
GI reflux (Gastrointestinal disorders) | 2
Heartburn (Dyspepsia) (Gastrointestinal disorders) | 7
Hemorrhage - vaginal (Reproductive system and breast disorders) | 2
Hypercalcemia (Metabolism and nutrition disorders) | 3
Hyperglycemia (Metabolism and nutrition disorders) | 12
Hypoalbuminemia (Metabolism and nutrition disorders) | 18
Hypocalcemia (Metabolism and nutrition disorders) | 12
Hypoglycemia (Metabolism and nutrition disorders) | 2
Hypokalemia (Metabolism and nutrition disorders) | 10
Hypomagnesemia (Metabolism and nutrition disorders) | 9
Hyponatremia (Metabolism and nutrition disorders) | 14
Insomnia (Psychiatric disorders) | 2
Leukocytopenia (Investigations) | 14
Lymphocyte count decreased (Investigations) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Nausea (Gastrointestinal disorders) | 10
Neutropenia (Investigations) | 7
Pelvic pain (Reproductive system and breast disorders) | 5
Peripheral limb edema (General disorders) | 4
Peripheral sensory neuropathy (Nervous system disorders) | 4
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2
Skin Ulceration (Skin and subcutaneous tissue disorders) | 2
Thrombocytopenia (Investigations) | 19
Urinary tract infection (Infections and infestations) | 4
Vomiting (Gastrointestinal disorders) | 5
Weight loss (Investigations) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less